CLINICAL TRIAL: NCT04011098
Title: Improving Labour Induction Analgesia: a Randomized Control Trial of Single Epidural Fentanyl Bolus at Epidural Initiation for Induction of Labour
Brief Title: Improving Labour Induction Analgesia: Epidural Fentanyl Bolus at Epidural Initiation for Induction of Labour
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Unable to meet recruitment numbers, lack of participation
Sponsor: University of Saskatchewan (Other)
Responsible Party: Principal Investigator, Harry Neveling, MD, University of Saskatchewan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Bio 18-73
Record Dates: First submitted 2019-06-06; First posted 2019-07-08 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Epidural; Labor Pain; Induction of Labor Affected Fetus / Newborn; Obstetric Anesthesia Problems; Obstetric Pain; Opioid
Keywords: Epidural; Opioids; Fentanyl; Labour Induction; Labour Pain; Obstetric Pain; Induction of Labour; Anesthesia; Obstetric Anesthesia
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Intervention Model Description: Prospective randomized control trial (RCT) utilizing parallel groups
Who Masked: Participant, Care Provider, Investigator
Masking Description: Participants will be randomized to one of two groups according to a 1:1 allocation with blinding of the intervention accomplished by providing the Anesthesia practitioner with either a 3 ml syringe filled with 2 ml of standard epidural mix (control) or 2 ml of Fentanyl (50 mcg/ml)(intervention):
  1. Control group: will receive a 2 ml bolus of standard epidural mix solution after epidural placement followed by standard care infusion of epidural local anesthetic/opioids, with a PCEA pump for subsequent analgesia.
  2. Fentanyl bolus group: will receive a 2 ml bolus of epidural Fentanyl (50 mcg/ml; therefore a total dose of 100 mcg) after epidural placement, followed by a standard care infusion of epidural local anesthetic/opioids, with a PCEA pump for subsequent analgesia.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Additional Epidural Fentanyl Bolus) (Active Comparator): The Control group will receive a 2 ml bolus of standard epidural mix solution after epidural placement followed by standard care infusion of epidural local anesthetic/opioids, with a PCEA pump for subsequent analgesia.
  Interventions: Drug: Standard Epidural Group
- Fentanyl bolus group (Experimental): The Fentanyl bolus group will receive a 2 ml bolus of epidural Fentanyl (50 mcg/ml; therefore a total dose of 100 mcg) after epidural placement, followed by a standard care infusion of epidural local anesthetic/opioids, with a PCEA pump for subsequent analgesia.
  Interventions: Drug: Epidural Fentanyl Bolus

INTERVENTIONS:
Drug: Epidural Fentanyl Bolus — Fentanyl bolus refers to the provision of a 2 ml bolus of epidural Fentanyl (50 mcg/ml; therefore a total dose of 100 mcg) after epidural placement, followed by a standard care infusion of epidural local anesthetic/opioids, with a PCEA pump for subsequent analgesia (0.08% Bupivicaine with 2 mcg/ml Fentanyl Solution).
  Other Names: Experimental Intervention
  Arms: Fentanyl bolus group
Drug: Standard Epidural Group — The Control group will receive a 2 ml bolus of standard epidural mix solution (0.08% Bupivicaine with 2 mcg/ml Fentanyl) after epidural placement followed by standard care infusion of the same solution, with a PCEA pump for subsequent analgesia.
  Other Names: Control Intervention
  Arms: Control Group (No Additional Epidural Fentanyl Bolus)

SUMMARY:
Labour pain can be intensified for labour inductions and women undergoing inductions often have earlier and more frequent requests for analgesia. Current evidence suggests that epidural analgesia effectively manages pain in labour, but may give rise to adverse effects for both the mother and neonate. Opioids are often added to epidurals to improve the quality of analgesia. Despite reassuring findings regarding epidural opioids, other investigators have found an association between epidural opioids and neonatal respiratory distress, lower Neurological and Adaptive Capacity scores, and reduced rates of breastfeeding. Given the heightened implications for the mother and neonate in situations requiring induction of labour, the desire for a positive outcome whilst still providing adequate maternal analgesia is paramount.

This study thus aims to investigate whether a preliminary epidural Fentanyl bolus at the initiation of the epidural may help to improve analgesia for women undergoing labour inductions for post-term pregnancy in a safe manner. Importantly, the main rationale of this proposed practice being that by achieving adequate epidural analgesia earlier in the labour induction, this may lead to better pain control overall and less overall requirements for epidural PCEA boluses and epidural "top-ups" as the induction progresses.

DETAILED DESCRIPTION:
The pain felt during labour is influenced by many physiological and psychosocial factors and often requires some form of relief. Pain can be intensified for labour inductions as the body's natural pain-relieving endorphins are not readily released in response to the increasingly strong and painful uterine contractions- leading to earlier and more frequent requests for analgesia. Induced labour has also been reported as being significantly longer than spontaneous labour. Current evidence suggests that epidural, combined spinal epidural and inhaled analgesia effectively manage pain in labour, but may give rise to adverse effects for both the mother and neonate. Despite this, epidural analgesia is considered the gold standard in the treatment of labor pain and has a role in labour inductions. Opioids are often added to epidurals to improve the quality of analgesia because of their faster onset and superior pain relief. When combined with opioids, lower concentrations of local anesthetic are needed. Such combinations provide adequate analgesic effect while allowing the parturient to maintain maximal motor function.

In studies assessing the safety and efficacy of labour analgesia, neonatal outcome is a primary concern and the use of opioids for labour analgesia is controversial because of the potentially negative effects on neonates. Common indicators of poor neonatal outcomes include a lower Apgar score, a lower Neurological and Adaptive Capacity Score (NACS), and a lower umbilical artery or vein pH value.

Fentanyl is the most widely investigated adjuncts to epidural local anesthetics. Various RCTs comparing epidural local anesthetics with and without fentanyl have found no significant differences in neonatal Apgar scores at one and five minutes between the groups. A recent meta-analysis of twenty-one RCTs involving epidural Fentanyl and Sufentanil concluded that there was no difference in the incidence of Apgar scores < 7 at one and five minutes, no significant differences in the NACS at two hours and at 24 hours, and no significant differences were found in umbilical cord artery pH between the epidural opioid and control groups. This meta-analysis concluded that the common doses of Fentanyl (total dose of 100-500 mcg) and Sufentanil (total dose of 7.5-30 mcg) used with an epidural/spinal technique are safe for neonates up to 24 hours after delivery. Despite reassuring findings regarding epidural opioids, other investigators have found an association between epidural opioids and neonatal respiratory distress and the use of epidural fentanyl has been associated with a NACS that failed to improve by 24 hours in one study. Furthermore, the use of epidural opioids was associated with reduced rates of breastfeeding in some observational studies, but evidence is unclear and debated.

Given the heightened implications for the mother and neonate in situations requiring induction of labour, the desire for a positive outcome whilst still providing adequate maternal analgesia is paramount. This study thus aims to investigate whether a preliminary epidural Fentanyl bolus at the initiation of the epidural may help to improve analgesia for women undergoing labour inductions for post-term pregnancy in a safe manner. Importantly, the main rationale of this proposed practice being that by achieving adequate epidural analgesia earlier in the labour induction, this may lead to better pain control overall and less overall requirements for epidural PCEA boluses and epidural "top-ups" as the induction progresses.

ELIGIBILITY:
Inclusion Criteria:

* Healthy parturients
* Parturients presenting for labour induction for post-term pregnancy (i.e. pregnancy beyond 42 weeks gestational age)
* Parturients who have had an uncomplicated pregnancy

Exclusion Criteria:

* Parturients presenting for induction of labour for pre-labour (premature) rupture of membranes
* Parturients presenting for induction of labour for hypertensive disorders of pregnancy [including preeclampsia, eclampsia, HELLP syndrome (Hemolysis, Elevated Liver enzymes, Low Platelets)]
* Parturients with maternal diabetes
* Fetal growth restriction
* Multiple gestation pregnancy
* Known or suspected Chorioamnionitis
* Known or suspected Abruptio placentae
* Oligohydramnios
* Parturients with cholestasis of pregnancy
* Known alloimmunization with fetal effects.
* Parturients with other chronic medical conditions or any complications related to pregnancy
* Participants who lack capacity to consent on their own behalf

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-11-02 (Actual); Study Completion 2020-11-02 (Actual)

PRIMARY OUTCOMES:
Labour analgesia quality: Change in verbal rating pain scale (VRS) after epidural placement | Verbal rating pain scale will be assessed 1) Prior to epidural placement, 2) 20 minutes after epidural placement, 3) 60 minutes after epidural placement, and 4) 120 minutes after epidural placement
  Quality of labour analgesia/pain scores will be assessed by the verbal rating pain scale (VRS) with a minimum score of 0 indicating "No Pain" and a maximum score of 10 indicating "Worst Possible Pain". Higher values closer to 10 indicate worse pain/poor analgesia. A score of 2 is indicative of "mild pain", a score of 4 is indicative of "moderate pain", a score of 6 is indicated of "severe pain", and a score of 8 is indicative of "very severe pain".
  Verbal rating pain scale will be assessed 1) Prior to epidural placement, 2) 20 minutes after epidural placement, 3) 60 minutes after epidural placement, and 4) 120 minutes after epidural placement.

SECONDARY OUTCOMES:
Total epidural opioid consumption | Total epidural opioid consumption will be summed following fetal delivery and discontinuation of the epidural infusion. The aim will be to collect this data within 24 hours of fetal delivery via chart review.
  Total opioid consumption will be measured by reviewing the epidural pump and adding together the total opioid infused and number PCEA or documented epidural "top-ups" or boluses.
Incidence of failed/incomplete epidurals | Incidence of failed/incomplete epidurals will be determined following fetal delivery and once all chart documents are available for review. The aim will be to collect this data within 24 hours of fetal delivery via chart review.
  Patient charts will be reviewed to look for any signs of a failed or incomplete/inadequate epidural (i.e. need to re-do epidural, concerns regarding incomplete block, need for multiple top-ups).
Neonatal well-being: Presence or Absence of Fetal Heart Tracing Abnormalities | Fetal Heart Tracing abnormalities will be assessed and summed following fetal delivery and once chart documents/fetal heart tracing strips are all available. The aim will be to collect this data within 24 hours of fetal delivery via chart review.
  Neonatal well-being will be assessed by monitoring for concerns charted about Fetal Heart Tracings. Specifically, patient charts will be reviewed to assess for concerns regarding early decelerations, late decelerations, and variable decelerations. The amount of decelerations will also be documented (if applicable).
Neonatal well-being: Apgar scores | Apgar scores will be recorded at 1 minute following fetal delivery and at 5 minutes following fetal delivery. The aim will be to collect this data within 24 hours of fetal delivery via chart review.
  Neonatal well-being will be assessed by recording Apgar scores at 1 minute following fetal delivery, and at 5 minutes following fetal delivery. The maximum and most reassuring Apgar score is 10 which indicates a neonate that is active, has a heart rate over 100 beats per minute, has a prompt response to stimulation, appears pink/well oxygenated and has a vigorous cry. In general, Apgar scores of 7 or higher are typically considered normal for a neonate and neonates with scores above 7 are unlikely to require resuscitative intervention.
  Any Apgar score below 7 is abnormal and should alert the care team of the possible need for resuscitative intervention. A score of 4-6 is below normal and means the neonate will likely need medical intervention or resuscitation. Apgar scores of 1-3 are critically low and indicative of a need for resuscitative intervention and intensive care.
Neonatal well-being: Umbilical artery pH value | Neonatal well-being will be assessed by recording the umbilical artery pH lab value at the time of fetal delivery/birth. The aim will be to collect this data within 24 hours of fetal delivery via chart review.
  Neonatal well-being will be assessed by recording and documenting the umbilical artery vein pH lab value drawn at the time of fetal delivery/birth. A umbilical artery pH value < 7.0 will be considered as abnormal and indicative of pathologic fetal acidemia.
Neonatal well-being: Breast-feeding quality | Neonatal breast-feeding quality will assessed and documented following fetal delivery and once all chart documents are available for review. The aim will be to collect this data within 48 hours of fetal delivery via chart review.
  Neonatal well-being will be assessed by reviewing postpartum patient charts to look for any documented consults to breastfeeding consultant (i.e. "yes" or "no" regarding the need for breastfeeding consultant). The number of breastfeeding consults will also be documented (if applicable).
Maternal well-being: Respiratory Rate | Maternal respiratory rate will be assessed 1) Prior to epidural placement, 2) Every 5 minutes after epidural placement until 20 minutes after epidural placement, 3) 60 minutes after epidural placement, and 4) 120 minutes after epidural placement
  Maternal well-being will be assessed by recording and documenting the maternal respiratory rate at specific intervals (see Time Frame below). A respiratory rate less than 12 will be considered as abnormal and bradypneic. A respiratory rate greater than 25 will be considered as abnormal and tachypneic.
Maternal well-being: Heart Rate | Maternal heart rate will be assessed 1) Prior to epidural placement, 2) Every 5 minutes after epidural placement until 20 minutes after epidural placement, 3) 60 minutes after epidural placement, and 4) 120 minutes after epidural placement
  Maternal well-being will be assessed by recording and documenting the maternal heart rate at specific intervals (see Time Frame below). A heart rate less than 60 beats per minute will be considered as abnormal and bradycardic. A heart rate greater than 110 beats per minute will be considered as abnormal and tachycardic.
Maternal well-being: Blood pressure | Maternal blood pressure will be assessed 1) Prior to epidural placement, 2) Every 5 minutes after epidural placement until 20 minutes after epidural placement, 3) 60 minutes after epidural placement, and 4) 120 minutes after epidural placement
  Maternal well-being will be assessed by recording and documenting the maternal blood pressure at specific intervals (see Time Frame below). Both systolic and diastolic blood pressures will be recorded. A systolic blood pressure less than 95 mmHg or a diastolic blood pressure less than 55 mmHg will be considered as abnormal and hypotensive. A systolic blood pressure greater than 140 mmHg or a diastolic blood pressure greater than 95 mmHg will be considered as abnormal and hypertensive.
Maternal well-being: Oxygen Saturation (SpO2) | Maternal oxygen saturation will be assessed 1) Prior to epidural placement, 2) Every 5 minutes after epidural placement until 20 minutes after epidural placement, 3) 60 minutes after epidural placement, and 4) 120 minutes after epidural placement
  Maternal well-being will be assessed by recording and documenting the maternal oxygen saturation at specific intervals (see Time Frame below). A maternal oxygen saturation less than 94% will be considered as abnormal and indicative of hypoxia.

CONTACTS AND LOCATIONS:
Overall Officials: Harry Neveling, MD, FRCPC, Principal Investigator — U of S Department of Anesthesiology, Perioperative Medicine and Pain Management
Locations (1):
- Royal University Hospital, Saskatoon, Saskatchewan, Canada

REFERENCES:
- [Background] Lowe NK. The nature of labor pain. Am J Obstet Gynecol. 2002 May;186(5 Suppl Nature):S16-24. doi: 10.1067/mob.2002.121427. PMID 12011870
- [Background] Simkin P, Bolding A. Update on nonpharmacologic approaches to relieve labor pain and prevent suffering. J Midwifery Womens Health. 2004 Nov-Dec;49(6):489-504. doi: 10.1016/j.jmwh.2004.07.007. PMID 15544978
- [Background] Melzack R. The myth of painless childbirth (the John J. Bonica lecture). Pain. 1984 Aug;19(4):321-337. doi: 10.1016/0304-3959(84)90079-4. No abstract available. PMID 6384895
- [Background] Poma S, Scudeller L, Gardella B, Broglia F, Ciceri M, Fuardo M, Pellicori S, Repossi F, Zizzi S, Noli S, Delmonte MP, Iotti GA. Outcomes of induced versus spontaneous labor. J Matern Fetal Neonatal Med. 2017 May;30(10):1133-1138. doi: 10.1080/14767058.2016.1205028. Epub 2016 Jul 13. PMID 27406914
- [Background] Rayburn WF. Minimizing the risks from elective induction of labor. J Reprod Med. 2007 Aug;52(8):671-6. PMID 17879826
- [Background] Jones L, Othman M, Dowswell T, Alfirevic Z, Gates S, Newburn M, Jordan S, Lavender T, Neilson JP. Pain management for women in labour: an overview of systematic reviews. Cochrane Database Syst Rev. 2012 Mar 14;2012(3):CD009234. doi: 10.1002/14651858.CD009234.pub2. PMID 22419342
- [Background] Wang K, Cao L, Deng Q, Sun LQ, Gu TY, Song J, Qi DY. The effects of epidural/spinal opioids in labour analgesia on neonatal outcomes: a meta-analysis of randomized controlled trials. Can J Anaesth. 2014 Aug;61(8):695-709. doi: 10.1007/s12630-014-0185-y. Epub 2014 Jul 11. PMID 25011701
- [Background] Anim-Somuah M, Smyth RM, Jones L. Epidural versus non-epidural or no analgesia in labour. Cochrane Database Syst Rev. 2011 Dec 7;(12):CD000331. doi: 10.1002/14651858.CD000331.pub3. PMID 22161362
- [Background] Russell R. The effects of regional analgesia on the progress of labour and delivery. Br J Anaesth. 2000 Jun;84(6):709-12. doi: 10.1093/bja/84.6.709. No abstract available. PMID 10895741
- [Background] Siddik-Sayyid SM, Taha SK, Azar MS, Hakki MA, Yaman RA, Baraka AS, Aouad MT. Comparison of three doses of epidural fentanyl followed by bupivacaine and fentanyl for labor analgesia. Acta Anaesthesiol Scand. 2008 Oct;52(9):1285-90. doi: 10.1111/j.1399-6576.2008.01765.x. PMID 18823470
- [Background] Beilin Y, Bodian CA, Weiser J, Hossain S, Arnold I, Feierman DE, Martin G, Holzman I. Effect of labor epidural analgesia with and without fentanyl on infant breast-feeding: a prospective, randomized, double-blind study. Anesthesiology. 2005 Dec;103(6):1211-7. doi: 10.1097/00000542-200512000-00016. PMID 16306734
- [Background] Nikkola EM, Jahnukainen TJ, Ekblad UU, Kero PO, Salonen MA. Neonatal monitoring after maternal fentanyl analgesia in labor. J Clin Monit Comput. 2000;16(8):597-608. doi: 10.1023/a:1012268617009. PMID 12580236
- [Background] Lee BB, Ngan Kee WD, Lau WM, Wong AS. Epidural infusions for labor analgesia: a comparison of 0.2% ropivacaine, 0.1% ropivacaine, and 0.1% ropivacaine with fentanyl. Reg Anesth Pain Med. 2002 Jan-Feb;27(1):31-6. doi: 10.1053/rapm.2002.27836. PMID 11799502
- [Background] Ruban P, Sia AT, Chong JL. The effect of adding fentanyl to ropivacaine 0.125% on patient-controlled epidural analgesia during labour. Anaesth Intensive Care. 2000 Oct;28(5):517-21. doi: 10.1177/0310057X0002800505. PMID 11094666
- [Background] Kumar M, Paes B. Epidural opioid analgesia and neonatal respiratory depression. J Perinatol. 2003 Jul-Aug;23(5):425-7. doi: 10.1038/sj.jp.7210905. PMID 12847541
- [Background] Loftus JR, Hill H, Cohen SE. Placental transfer and neonatal effects of epidural sufentanil and fentanyl administered with bupivacaine during labor. Anesthesiology. 1995 Aug;83(2):300-8. doi: 10.1097/00000542-199508000-00010. PMID 7631952
- [Background] Jordan S, Emery S, Bradshaw C, Watkins A, Friswell W. The impact of intrapartum analgesia on infant feeding. BJOG. 2005 Jul;112(7):927-34. doi: 10.1111/j.1471-0528.2005.00548.x. PMID 15957994
- [Background] Torvaldsen S, Roberts CL, Simpson JM, Thompson JF, Ellwood DA. Intrapartum epidural analgesia and breastfeeding: a prospective cohort study. Int Breastfeed J. 2006 Dec 11;1:24. doi: 10.1186/1746-4358-1-24. PMID 17134489
- [Background] Reynolds F. Labour analgesia and the baby: good news is no news. Int J Obstet Anesth. 2011 Jan;20(1):38-50. doi: 10.1016/j.ijoa.2010.08.004. Epub 2010 Dec 13. PMID 21146977
- [Background] Wilson MJ, MacArthur C, Cooper GM, Bick D, Moore PA, Shennan A; COMET Study Group UK. Epidural analgesia and breastfeeding: a randomised controlled trial of epidural techniques with and without fentanyl and a non-epidural comparison group. Anaesthesia. 2010 Feb;65(2):145-53. doi: 10.1111/j.1365-2044.2009.06136.x. Epub 2009 Nov 12. PMID 19912160